CLINICAL TRIAL: NCT04815317
Title: Sensory and Emotional Modulation of Dyspnea Under Artificial Ventilation in the Intensive Care Unit
Acronym: Sensopnée2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Association pour le Développement et l'Organisation de la Recherche en Pneumologie et sur le Sommeil (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 2019-A01532-55
Record Dates: First submitted 2021-02-10; First posted 2021-03-25 (Actual); Last update posted 2022-09-02 (Actual); Status verified 2022-01

CONDITIONS: Dyspnea
Keywords: Patient-ventilator interaction; Inspiratory muscles; Electromyogram; Mechanical ventilation
MeSH Terms: conditions — Dyspnea | interventions — Sensitive Tartar Control Dentifrice

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Basal (Active Comparator): The impact of these stimulations will be compared to that of a control stimulus.
  The auditory control condition will consist of listening to a pink noise. The pink noise, like the white noise, is a normalized noise. The sound produced on a TV set that is out of adjustment during the "snow effect" is a representative example of such noise. Pink noise is a random signal whose power spectral density decreases by 3dB per octave. This signal is closer to the sensitivity of the ear than white noise.
  The sensitive control condition will be achieved by administering fresh air on the calf.
  An pressure support (+5) increment will be performed to ensure comparability of subsequent experimental sequences and their effect on dyspnea.
  Interventions: Other: Auditory control; Other: Sensitive control
- Intervention (Experimental): Patients will be subjected to sensory stimuli that may be auditory or sensitive.
  The sensory stimulations will be administered by a research nurse. The auditory stimulation will consist of listening to relaxing pieces of music from MP3 files from the International Center for Music Therapy (Noisy le Grand, France).
  Listening will be done through noise-cancelling headphones (PLANTRONICS, Gamecom 780, Santa Cruz, California, USA) for 10 minutes.
  Sensitive stimulation will consist of administering fresh air to the patient's face by means of a fan without blades (DYSON AM01, Malmesbury, UK) for 10 minutes.
  Interventions: Other: Auditive stimulation; Other: Sensitive stimulation

INTERVENTIONS:
Other: Auditive stimulation — The auditory stimulation will consist of listening to relaxing pieces of music from MP3 files from the International Center for Music Therapy (Noisy le Grand, France).
  Listening will be done through noise-cancelling headphones (PLANTRONICS, Gamecom 780, Santa Cruz, California, USA) for 10 minutes.
  Arms: Intervention
Other: Sensitive stimulation — Sensitive stimulation will consist of administering fresh air to the patient's face by means of a fan without blades (DYSON AM01, Malmesbury, UK) for 10 minutes.
  Arms: Intervention
Other: Auditory control — The auditory control condition will consist of listening to a pink noise. The pink noise, like the white noise, is a normalized noise. The sound produced on a TV set that is out of adjustment during the "snow effect" is a representative example of such noise. Pink noise is a random signal whose power spectral density decreases by 3dB per octave. This signal is closer to the sensitivity of the ear than white noise.
  Arms: Basal
Other: Sensitive control — The sensitive control condition will be achieved by administering fresh air on the calf.
  Arms: Basal

SUMMARY:
Rationale: Half of the patients receiving mechanical ventilation in the intensive care unit (ICU) have moderate to severe dyspnea. This dyspnea has a negative impact on the duration of mechanical ventilation, on patients' comfort and could be involved in the genesis of post-traumatic stress syndromes, a frequent complication of intensive care. Modifying ventilation parameters does not always relieve dyspnea and administering morphine prolongs the duration of mechanical ventilation. Dyspnea has, in addition to its sensory component, an emotional component. The possibility to distract the patients' attention or to modulate their emotions in order to relieve their dyspnea could therefore represent an innovative therapeutic alternative devoid of side effects.

Objectives: To evaluate the effect of auditory and sensory extra respiratory stimuli on the sensation of dyspnea in intensive care patients undergoing mechanical, invasive or non-invasive ventilation.

Methods: 45 intensive care patients under artificial ventilation will be exposed, according to their randomization arm, to the following two stimuli for a duration of 10 minutes:

* standard relaxing music piece versus "pink" noise;
* fresh air on the face versus fresh air on the thigh. The effect of this stimulus will be compared to a randomized control, these two conditions will be separated by a wash-out period.

An pressure support (+5) increment will be performed to ensure comparability of subsequent experimental sequences and their effect on dyspnea.

Dyspnea will be assessed in terms of intensity (visual analog scale) and characterized sensorially. Will also be evaluated during the different conditions: pain, anxiety and stress (sympathetic/parasympathetic balance) and extra-diaphragmatic electromyographic activity.

Ethical framework: research involving the human person at risk and minimal constraints (physiology study that does not entail any risk for the patients).

Expected results and prospects: the investigators hypothesize that pleasant extra-respiratory sensory stimulation significantly reduces the intensity of dyspnea in artificially ventilated patients without any change in ventilator settings and pharmacological intervention. This reduction in dyspnea is associated with decreased anxiety and stress levels.

This study will bring new, easy-to-use and side-effect-free tools to the therapeutic arsenal for the relief of dyspnea in mechanically ventilated patients.

DETAILED DESCRIPTION:
Dyspnea or "shortness of breath" is a major symptom that alters the quality of life of patients who suffer from it. It is a multimodal sensation that integrates psychological, social and environmental factors (1). Recent studies have shown that dyspnea and pain share a number of characteristics (2). In intensive care, dyspnea affects up to half of the patients under mechanical ventilation (3). However, unlike pain, which has been the subject of numerous studies in intensive care, relieving it is not a usual therapeutic objective.

In recent years, despite considerable progress in the understanding of the mechanisms of dyspnea, there has been no major advance in the therapeutic tools aimed at relieving it. The best evaluated and most prescribed drugs currently available to relieve dyspnea are morphine drugs (4). However, there is no formal proof of their long-term effectiveness and side effects such as the respiratory depressant effect make them difficult to use. Non-pharmacological tools integrating the sensory but also emotional dimension of dyspnea have also been developed. The investigators find parallel medicines (acupuncture, hypnosis...) but also extra respiratory stimulation techniques (thoracic vibrations, administration of fresh air to the face...) which modulate and relieve dyspnea with a certain success (1).

Optimizing tools to relieve dyspnea patients is therefore a priority. To date, the pharmacological arsenal is limited due to the number of effective molecules and their side effects. Non-pharmacological tools allowing to modulate the sensory and emotional components of dyspnea represent a therapeutic alternative that deserves to be explored. This is the purpose of this project.

Half of the patients undergoing mechanical ventilation in intensive care have moderate to severe dyspnea. This dyspnea has a negative impact on the duration of mechanical ventilation, on patient comfort and on the incidence of post-traumatic stress disorder. Changing ventilation parameters does not always relieve dyspnea, and administering morphine prolongs the duration of mechanical ventilation. The possibility of distracting the patients' attention or modulating their emotions in order to relieve their dyspnea seems to be a simple way to improve their comfort and could represent an innovative therapeutic alternative.

In this context, the investigators hypothesize that pleasant extra respiratory sensory stimulation relieves dyspnea in artificially ventilated patients without any change in ventilator settings and pharmacological intervention.

The main objective of our study is to demonstrate, in dyspneic patients undergoing artificial ventilation, a decrease in dyspnea under the effect of :

* listening to a piece of music versus pink noise;
* the application of cold air to the face versus the application of cold air to the calf.

The secondary objectives are to evaluate the effect of extra-respiratory stimuli on :

* the quality of dyspnea (thirst for air, excessive respiratory work, concentration)
* the intensity of secondary emotional responses (anxiety, fear).
* the electromyographic activity of extra-diaphragmatic inspiratory muscles

STUDY CONDITIONS The experimental sessions will take place in the patient's room, in the Intensive Care Unit of Prof. T. Similowski.

Patients will have been previously informed orally and in writing and will have signed the informed consent.

TYPE OF STUDY It is research involving the human person with minimal risk and constraints, interventional, open, randomized.

POPULATION, SAMPLING All subjects, without exception, must understand French and have read and understood the appropriate information leaflet and signed the consent form.

It is research involving the human person with minimal risk and constraints, interventional, open, randomized.

PATIENT MONITORING During the experimental sessions, an investigating physician will systematically be present in the room. Any tolerance abnormality (agitation, disturbance of vigilance, SpO2 <88%, tachycardia greater than 130/min or mean blood pressure < 60mmHG) will lead to the interruption of the experimental session.

EXPERIMENTAL PROTOCOL Each patient will participate in a single one-hour experimental session that will take place as follows.

The type of stimulation administered to the patient will be determined by randomization. The order of administration of the stimulation and its control will also be determined by randomization.

Each experimental session will consist of ten sequences of 10 minutes each.

The experimental sequences will proceed as follows:

BASIC: recording of ventilation parameters, constants, ECG, skin conductance and psycho-sensory parameters at baseline.

PRESSURE SUPPORT INCREMENT: An pressure support (+5) increment will be performed to ensure comparability of subsequent experimental sequences and their effect on dyspnea.

WASH OUT: new recording in basic ventilation. Sensory and psycho-sensory parameters are again collected as above.

STIMULUS 1 case or control: administration of extra-respiratory stimulation 1 or its control depending on the randomization arm. Sensory and psycho-sensory variables are measured as above.

WASH OUT: new recording in basic ventilation. Sensory and psycho-sensory parameters are again collected as above.

STIMULUS 1 case or control: administration of extra-respiratory stimulation 1 or its control according to the randomization arm. Sensory and psycho-sensory variables are measured as above.

WASH OUT: new recording in basic ventilation. Sensory and psycho-sensory parameters are again collected as above.

STIMULUS 2 cases or control: administration of extra respiratory stimulation 1 or its control according to the randomization arm. Sensory and psycho-sensory variables are measured as above.

WASH OUT: new recording in basic ventilation. Sensory and psycho-sensory parameters are again collected as above.

STIMULUS 2 cases or control: administration of extra respiratory stimulation 1 or its control according to the randomization arm. Sensory and psycho-sensory variables are measured as above.

RECOVERY: Interruption of the stimulation or its control is interrupted. Recording of ventilatory, sensory and psycho-sensory parameters after return to baseline.

ELIGIBILITY:
Inclusion Criteria:

* Mechanical ventilation : invasive for at least 48 hours or non-invasive for at least 24 hours, sequential or continuous
* Dyspnea ≥ 4 on a visual analogic scale (VAS) from 0 to 10
* Absence of delirium (evaluated by the CAM-ICU score) ;
* Communicative patient

Exclusion Criteria:

* Patients on ECMO or decarboxylation ;
* Patients on long-term left ventricular support;
* Patients postoperatively following any surgery (pain from the procedure may interfere with dyspnea);
* Protected minors and adults;
* Pregnant women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2019-11-26 (Actual); Primary Completion 2021-08-27 (Actual); Study Completion 2021-11-26 (Actual)

PRIMARY OUTCOMES:
Detection and quantification of dyspnea intensity change | At the baseline and during the interventions
  Dyspnea will initially be searched for with absence or presence. If present, it will then be quantified using a visual analog scale graduated from 0 ("absence of respiratory discomfort") to 10 ("maximum respiratory discomfort").

SECONDARY OUTCOMES:
Anxiety | At the baseline and during the interventions
  Anxiety will be sought initially. If it is present, it will then be evaluated using a visual analog scale graduated from 0 ("absence of anxiety") to 10 ("maximum anxiety").
Mesure of pain | At the baseline and during the interventions
  Patients in resuscitation can be painful, which can interfere with the perception of dyspnea. Pain will be sought first.If it is present, it will then be assessed using a visual analogue scale graduated from 0 ("no pain") to 10 ("maximum pain").
  Discomfort caused by the stimulus The inconvenience caused by the stimuli applied to the patient will be quantified, if any, using a visual analog scale graduated from 0 ("no inconvenience") to 10 ("maximum inconvenience").
Electromyogram of extra-diaphragmatic inspiratory muscles | At the baseline and during the interventions
  Electromyogram (EMG) of the extra-diaphragmatic inspiratory muscles: the amplitude of the EMG signal of the extra-diaphragmatic inspiratory muscles is proportional to the intensity of the dyspnea. It will be collected by self-adhesive surface electrodes of the same type as those usually used to collect the ECG signal in intensive care patients. A distance of 2 cm will separate the two electrodes. The position of the electrodes will depend on the muscle whose EMG activity is collected: scalene muscles, intercostal parasternal muscles, Alae nasi muscles, etc. The EMG signal will be amplified (PowerLab, AD Instruments, Hastings, UK), then sampled at a frequency of 10 kHz and finally filtered between 40 and 500 Hz.

CONTACTS AND LOCATIONS:
Overall Officials: Alexandre DEMOULE, MD, PhD, Principal Investigator — Groupe Hospitalier Universitaire APHP - Sorbonne Université Site Pitié-Salpêtrière (bâtiment Eole)
Locations (1):
- Service de Pneumologie et Réanimation Médicale, Groupe Hospitalier Pitié Salpêtrière, Paris, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Parshall MB, Schwartzstein RM, Adams L, Banzett RB, Manning HL, Bourbeau J, Calverley PM, Gift AG, Harver A, Lareau SC, Mahler DA, Meek PM, O'Donnell DE; American Thoracic Society Committee on Dyspnea. An official American Thoracic Society statement: update on the mechanisms, assessment, and management of dyspnea. Am J Respir Crit Care Med. 2012 Feb 15;185(4):435-52. doi: 10.1164/rccm.201111-2042ST. PMID 22336677
- [Background] Morelot-Panzini C, Demoule A, Straus C, Zelter M, Derenne JP, Willer JC, Similowski T. Dyspnea as a noxious sensation: inspiratory threshold loading may trigger diffuse noxious inhibitory controls in humans. J Neurophysiol. 2007 Feb;97(2):1396-404. doi: 10.1152/jn.00116.2006. Epub 2006 Jul 26. PMID 16870842
- [Background] Schmidt M, Demoule A, Polito A, Porchet R, Aboab J, Siami S, Morelot-Panzini C, Similowski T, Sharshar T. Dyspnea in mechanically ventilated critically ill patients. Crit Care Med. 2011 Sep;39(9):2059-65. doi: 10.1097/CCM.0b013e31821e8779. PMID 21572329
- [Background] Abernethy AP, Currow DC, Frith P, Fazekas BS, McHugh A, Bui C. Randomised, double blind, placebo controlled crossover trial of sustained release morphine for the management of refractory dyspnoea. BMJ. 2003 Sep 6;327(7414):523-8. doi: 10.1136/bmj.327.7414.523. PMID 12958109
- [Background] Lansing RW, Gracely RH, Banzett RB. The multiple dimensions of dyspnea: review and hypotheses. Respir Physiol Neurobiol. 2009 May 30;167(1):53-60. doi: 10.1016/j.resp.2008.07.012. Epub 2008 Jul 25. PMID 18706531